CLINICAL TRIAL: NCT02626442
Title: Exercise and Brain Health
Acronym: EBH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baltimore VA Medical Center (U.S. Federal Agency)
Collaborators: University of Maryland (Other)
Responsible Party: Principal Investigator, Rich Macko, Associate Director of Research for the GRECC, Baltimore VA Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BaltimoreVAMC
Record Dates: First submitted 2015-11-18; First posted 2015-12-10 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Stroke; Cardiovascular Risk Factors; Transient Ischemic Attack (TIA)
Keywords: Cognition; Exercise
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group Exercise Class (Experimental): 6 month group balance/exercise class, three days a week - up to one hour. Exercise program includes walking around a track, bodyweight/balance exercises, and an obstacle course.
  Interventions: Other: Exercise
- Testing (No Intervention): Subjects enrolled in other MERCE exercise and robotics interventions will receive balance/walking tests, MRI with famous name recognition task, and cognitive testing pre and post their intervention.

INTERVENTIONS:
Other: Exercise — 6 month group exercise class
  Arms: Group Exercise Class

SUMMARY:
The risk of stroke and vascular dementia is high in individuals who have had a prior stroke or TIA, and in those who have vascular disease risk factors, such as high blood pressure, abnormal cholesterol, diabetes or pre-diabetes. These vascular risk factors can improve with exercise. This study will examine the impact of a 6 month, low intensity group exercise class on fitness, walking, balance, and brain health.

This study will also collect fitness, walking, balance, and brain health outcome measures at baseline and post all other MERCE exercise and robotics interventions.

DETAILED DESCRIPTION:
A major public health problem in aging is that about half of all stroke survivors have significant cognitive problems, called vascular cognitive impairment, nondementia (VCIND) and also a 10fold increased risk of going on to develop full dementia. Investigators at University of Maryland and VA Maryland Exercise and Robotics Center of Excellence (MERCE) have developed exercise programs for individuals that have suffered a disabling stroke that improve cardiovascular fitness levels, walking function, balance, and can reverse impaired glucose tolerance (prediabetic state) and non-insulin dependent diabetes in nearly 60% of stroke patients. Our most recent randomized studies provide the first evidence that aerobic exercise (cardiovascular) can improve selected aspects of cognitive function that typically decline with aging, and can increase indirect measures of blood flow to the brain. All of these findings provide hope that exercise can improve brain health by reducing recurrent stroke including silent strokes (9/10 stroke are silent), and improving cognitive function. Yet, no studies to our knowledge have shown that exercise training can improve these elements of brain health in individuals that have had a minor stroke, silent strokes, or are at great risk of stroke due to the presence of cerebrovascular risk factors (e.g., hypertension, prediabetes, etc.). Research studies in this pilot clinical demonstration project are designed to: 1) provide new insights into the potential role for exercise to improve brain health in aging and after minor stroke or at risk for stroke by using advanced brain imaging techniques; 2) extend our findings in exercise and brain health to a population with cerebrovascular disease, including those with less severe neurological deficits; those with cerebrovascular risk factors, minor strokes, transient ischemic attack (neurological deficits resolved, but still at high risk for further events), or silent strokes, which are extremely common and predictive of developing cognitive decline and dementia. Furthermore, the investigators are dedicated to testing exercise programs that can reach out to the community. Therefore, the investigators propose to use the same low intensity exercise class format that the investigators already have implemented safely and effectively at County Senior Centers in Maryland over the last 4 years for more disabled stroke patients, toward the training of these minimally disabled or nondisabled older individuals with silent or minor cerebrovascular disease. The results of this study will lay the groundwork for community partnering and broader dissemination providing exercise programs designed to preserve and improve brain health for those at high risk of vascular disease and cognitive decline in aging. The hypothesis is that a 6 month supervised exercise class will improve brain function and cognitive function among individuals with cerebrovascular risk factors, minor stroke, TIA, or silent stroke as indicated by measures before and after training of 1) written and computer - based cognitive function (memory and thinking) and mood tests and 2) MRI pictures of the brain to see if blood flow is increased or damage due to old strokes and aging is reduced by the exercise training.

Individuals with cerebrovascular risk factors (e.g., hypertension, diabetes), minor stroke (nondisabling stroke in terms of community or home walking capability), TIA (warning stroke), or silent stroke (seen by brain imaging, but no paralysis or obvious stroke signs or symptoms) will be entered into a 6 month duration exercise class.

Initial medical and neurological evaluation will be conducted by a credentialed Clinician to assure that individuals are eligible and that they are medically and neurologically approved for participation in a low intensity aerobic exercise class. All subjects will have approval of their primary care provider, documenting their awareness and medical approval for their patient to enter into a low to moderate exercise intensity class. This is the same medical clearance that is already Institutional Review Board approved and is in use for the similar exercise class for stroke and neurologic disability in Howard County Department of Aging Senior Centers. Before starting the exercise, all subjects will be given a series of baseline testing: 1) walking and balance tests to characterize their mobility performance capacity (timed walks, Short Physical Performance Battery, Functional Reach, Berg Balance Test, modified dynamic gait index, and 4 square stepping, 2) a 12 hour battery of written and computer based cognitive function and mood tests and questionnaires, and 3) MRI that lasts about 1 hour that includes pictures of the brain . All of these tests will be repeated at midpoints (i.e., 3 months) and at the end of the training program (6 months, MRIs are performed only at baseline and 6 months). The exercise class will consist of supervised walking as well as bar and chair exercises to address upper and lower extremity function. The class will occur 3 times per week for 6 months.

Individuals are instructed to perform select parallel exercises at home the remaining days of the weeks and record activities in a homework logbook.

This protocol is being designed in a modular fashion to collect the same outcomes at baseline and post all other MERCE exercise and robotics interventions.

ELIGIBILITY:
Inclusion Criteria:

* Adequate language and neurocognitive function to participate in testing and training and to give adequate informed consent
* Able to rise from a chair unaided
* Completion of all regular post-stroke physical therapy (if applicable)
* Able to walk 30 feet without human assistance

Exclusion Criteria:

* Clinical history of

  * unstable angina
  * recent (< 3 months) myocardial infarction or congestive heart failure (NYHA category II)
  * hemodynamically significant valvular dysfunction
  * peripheral arterial obstructive disorder with claudication
  * major orthopedic, chronic pain, or non-stroke neuromuscular disorders restricting exercise
  * pulmonary or renal failure
  * poorly controlled hypertension (>190/110), measured on at least two separate occasions
  * recent hospitalization for severe disease or surgery
  * severe or global receptive aphasia which confounds reliable testing and training
  * Other medical condition precluding patient participation in this study as per medical judgment of study team
* Untreated major depression
* Pregnancy
* Alcohol consumption > 3 oz. liquor, or 3 x 4 oz glasses of wine, or 3 x 12 oz. beers per day, by self-report
* Dementia and other major cognitive deficits (based upon clinical evaluation)

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2013-07; Primary Completion 2020-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in executive function | 6 months
  Measured by cognitive battery
Change from baseline in cortical thickness | 6 month
  Measured during brain MRI
Change from baseline in EEG | 6 month
  EEG will be performed during tasks
Change from baseline in hippocampal volume | 6 month
  Measured during brain MRI

CONTACTS AND LOCATIONS:
Overall Officials: Emily Byrne, BS, Study Director — Baltimore VA Medical Center
Locations (1):
- Baltimore VA Medical Center, Baltimore, Maryland, United States